CLINICAL TRIAL: NCT02392338
Title: Comparison of Success Rate of Totally Thoracoscopic Ablation Versus Hybrid Procedure in Patients With Persistent Atrial Fibrillation
Brief Title: Hybrid Procedure in Patients With Persistent Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Young Keun On, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-10-090
Record Dates: First submitted 2014-11-10; First posted 2015-03-19 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Ablation; Hybrid
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Thoracoscopic ablation group (No Intervention): Patients who will undergo thoracoscopic ablation only
- Hybrid procedure (Active Comparator): Patients who will undergo hybrid procedure (thoracoscopic ablation and eletrophyologic study with or without additional ablation)
  Interventions: Procedure: Hybrid procedure

INTERVENTIONS:
Procedure: Hybrid procedure — Eletrophysiologic study via femoral vein approach to confirm pulmonary vein isolation lesion and box lesions in left atrium
  Other Names: Postprocedural electrophysiological study
  Arms: Hybrid procedure

SUMMARY:
In this study, the investigators therefore comparatively analyzed the mid-term results (at 1 year) including electrocardiogram, 24 hour Holter monitoring, and 2 week long-term electrocardiogram of thoracoscopic ablation and RFCA performed individually or as a hybrid procedure in patients with long-lasting persistent atrial fibrillation. Antiarrhythmic medication, discontinuation of anticoagulation medication, and echocardiographic findings were also analyzed.

DETAILED DESCRIPTION:
Atrial fibrillation is highly associated with sudden death and stroke, requiring definitive treatment. In Korea, atrial fibrillation is a common disease predicted to affect more than 5% of the population over 65 years of age and more than 10% over 80 years.

Totally thoracoscopic ablation has been adopted and performed successfully on February 2012 at Samsung Medical Center for the first time in Korea. More than 120 operations have been performed up to date.

In Korea, treatment for atrial fibrillation is still dependent on percutaneous RFCA, and life-long medication and anticoagulation is needed when recurrent atrial fibrillation occurs. The investigators expected thoracoscopic ablation to be an alternative to overcome this limitation. Also, thoracoscopic ablation and RFCA are recently being performed simultaneously or stage by stage as a hybrid procedure, and the results are being reported.

In this study, the investigators therefore comparatively analyzed the mid-term results (at 1 year) including electrocardiogram and 24 hour Holter monitoring of thoracoscopic ablation and RFCA performed individually or as a hybrid procedure in patients with long-lasting persistent atrial fibrillation. Antiarrhythmic medication, discontinuation of anticoagulation medication, and echocardiographic findings were also analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Long-lasting persistent atrial fibrillation
2. Persistent atrial fibrillation refractory to antiarrhythmic drug therapy
3. over 18 years

Exclusion Criteria:

1. Valvular heart disease of more than moderate degree
2. Unresponsive ischemic cardiomyopathy
3. Follow-up of over 1 year was not possible
4. Warfarin was unable to be used
5. Refusal of informed consent
6. Left atrial thrombus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-11; Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Cardiac related death | one year
  medical records review

SECONDARY OUTCOMES:
Stroke | postoperative one year
  medical records review at 3, 6 and 12 months follow up
Bleeding | postoperative one year
  medical records review at 3, 6 and 12 months follow up
Embolism | postoperative one year
  medical records review at 3, 6 and 12 months follow up
Recurred atrial arrhythmia | postoperative one year
  medical records review at 3, 6 and 12 months follow up

CONTACTS AND LOCATIONS:
Overall Officials: Young Keun On, MD,PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pison L, La Meir M, van Opstal J, Blaauw Y, Maessen J, Crijns HJ. Hybrid thoracoscopic surgical and transvenous catheter ablation of atrial fibrillation. J Am Coll Cardiol. 2012 Jul 3;60(1):54-61. doi: 10.1016/j.jacc.2011.12.055. PMID 22742400
- [Derived] Choi MS, On YK, Jeong DS, Park KM, Park SJ, Kim JS, Carriere KC. Usefulness of Postprocedural Electrophysiological Confirmation Upon Totally Thoracoscopic Ablation in Persistent Atrial Fibrillation. Am J Cardiol. 2020 Apr 1;125(7):1054-1062. doi: 10.1016/j.amjcard.2019.12.046. Epub 2020 Jan 8. PMID 31948665